CLINICAL TRIAL: NCT05500326
Title: Ivermectin Therapy for Scabies Infection in Children Younger Than 5 Years of Age (ITCHY Study)
Acronym: ITCHY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Burnet Institute (Other); Lao Tropical and Public Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 84086
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-02

CONDITIONS: Scabies; Itch; Scabies
Keywords: Neglected tropical diseases
MeSH Terms: conditions — Scabies; Pruritus; Neglected Diseases | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): ITCHY Study:
  All participants will receive one dose of oral 3mg Ivermectin tablet.
  ITCHY2 study:
  Participants will receive one age-specific dose of oral ivermectin tablet.
  Age specific ivermectin dose:
  * 0.75mg of ivermectin will be given to participants aged 3 to 7 months
  * 1.5mg of ivermectin will be given to participants aged 8 to 12 months
  * 3mg of ivermectin will be given to participants aged 13 to 24 months
  Interventions: Drug: Ivermectin Tablets

INTERVENTIONS:
Drug: Ivermectin Tablets — ITCHY Study:
  All participants will receive one dose of oral ivermectin 3mg on day 0 and have two blood samples taken to determine the serum ivermectin concentrations after the dose. Timing of blood samples will vary depending on the allocated group.
  ITCHY2 Study:
  Participants will receive one age-specific dose of oral ivermectin on day 0 and have two blood samples taken to determine the serum ivermectin concentrations after the dose. Timing of blood samples will vary depending on the allocated group.
  Age specific ivermectin dose:
  * 0.75mg of ivermectin will be given to participants aged 3 to 7 months
  * 1.5mg of ivermectin will be given to participants aged 8 to 12 months
  * 3mg of ivermectin will be given to participants aged 13 to 24 months

SUMMARY:
This is an open label prospective pharmacokinetic single arm study in Laos PDR. This study will be embedded within a cluster-randomized controlled trial of interventions to address childhood undernutrition (SUANHOAM Trial, ACTRN12620000520932) and involves a collaboration with the Murdoch Children's Research Institute, Burnet institute and Lao Tropical and Public Health Institute.

ITCHY Study:

The primary objective is to determine in young children aged 2 to <5 years and weighing 10 to <15 kg if an ivermectin dose of 3 mg achieves comparable drug exposures to the recommended dose in older children. It aims to provide reliable evidence for a safe and effective dose of ivermectin in young children who are especially vulnerable to scabies infections and the associated secondary complications.

ITCHY2 Study:

An embedded phase 2 multicentre, open label prospective pharmacokinetic study in Laos PDR of ITCHY Study. The primary objective is to determine the plasma ivermectin drug exposure in children aged 3 months to 2 years and weighing ≥2 kg receiving an age specific ivermectin dose.

DETAILED DESCRIPTION:
ITCHY study:

100 children aged 2 to <5years and weighing 10 to <15 kg with clinically diagnosed scabies infection in the participating sites in Laos PDR will be approached for recruitment into the study if eligible (see eligibility criteria) and allocated into one of four blood sampling groups with 25 participants in each group. The 3mg dose of ivermectin will be administered orally and blood samples will be collected at two different time points accordingly to blood sampling groups allocation after the first 3mg dose of ivermectin. Clinical responses will be assessed on day 14. A second dose of ivermectin to complete the treatment will only be administered if the first dose has been tolerated by the participants. The 3mg ivermectin drug exposure, safety and effectiveness will be measured.

ITCHY2 Study:

120 children aged 3 months to 2 years and weighing ≥2 kg with clinically diagnosed scabies infection in the participating sites in Laos PDR will be approached for recruitment into the study if eligible (see eligibility criteria) and allocated into one of four blood sampling groups with 30 participants in each group. An age specific dose of ivermectin will be administered orally and blood samples will be collected at two different time points accordingly to blood sampling groups allocation after the first dose of ivermectin.

Age specific ivermectin dose:

* 0.75mg of ivermectin will be given to participants aged 3 to 7 months
* 1.5mg of ivermectin will be given to participants aged 8 to 12 months
* 3mg of ivermectin will be given to participants aged 13 to 24 months

Clinical responses of the participants will be assessed on day 14. A second age specific dose of ivermectin to complete the treatment will only be administered if the first dose has been tolerated by the participants. The ivermectin plasma drug exposure, safety and effectiveness will be measured.

ELIGIBILITY:
Inclusion Criteria

ITCHY study:

Children aged 2 to <5 years and weighing 10 to <15 kg with scabies infection as clinically diagnosed by the treating clinician.

ITCHY2 study:

Children aged 3 months to 2 years and weighing ≥2 kg with scabies infection as clinically diagnosed by the treating clinician.

Exclusion Criteria:

ITCHY and ITCHY2 study:

* Children with known liver disease
* Children with known allergy to ivermectin
* Children with concomitant warfarin use
* Children with known neurological disease
* Children already receiving topical treatment for scabies

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ivermectin drug exposure - Area under the concentration-time curve (AUC0- ∞ ) | ITCHY study: 20minutes, 2 hours, 6 hours, 12 hours, 24 hours, 48 hours and 96 hours post-dose. ITCHY2 study: 90mins, 5 hours, 6 hours, 12 hours, 24 hours, 48 hours and 96 hours post dose.
  ITCHY study:
  * The mean (standard deviation) of ivermectin exposure as measured by the area under the concentration-time curve (AUC0) in the study population of children aged 2 to <5 years and weighing 10 to <15 kg. The calculated AUC will be AUC0- ∞ i.e. from time 0 extrapolated to infinity for a single dose.
  * Comparable drug exposure will be defined as the mean ivermectin AUC in the study population being ≥80% (efficacy boundary) and ≤125% (toxicity boundary) of the mean AUC in the children aged ≥5 years and weighing ≥15 kg from our previous study with 90% confidence Intervals.
  ITCHY2 study:
  -The mean (standard deviation) plasma ivermectin exposure as measured by the area under the concentration-time curve (AUC0-∞) after the first ivermectin dose in the study population of children aged 3 months to 2 years and weighing ≥2 kg. The calculated AUC will be AUC0-∞ i.e. from time 0 extrapolated to infinity for a single dose.

SECONDARY OUTCOMES:
Proportion of participants with at least one ivermectin-related adverse event | Post intervention at Day 14
  ITCHY and ITCHY2 study: Causality will be assessed using the Naranjo Adverse Drug Reaction Probability Scale Worksheet. The Naranjo Algorithm, or Adverse Drug Reaction Probability Scale, is a method by which to assess whether there is a causal relationship between an identified untoward clinical event and a drug using a questionnaire to assign probability scores.
The proportion of participants whose scabies infection has improved after treatment with ivermectin | Day 0 and post-intervention at Day 14
  ITCHY and ITCHY2 study: The proportion of children whose scabies infection has improved at 14 days as assessed by the same treating clinician as on day 0. The severity of scabies infection will be measured using a descriptive scale (No Change, Improved -Completely resolved, improved-partially resolved, worsened, other, unknown) , the outcome will be presented as descriptive data (i.e percentage of participants in each category of the scale )

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gwee, PhD, Principal Investigator — Murdoch Childrens Research Institute (MCRI)
Locations (5):
- Laos (5):
  - Banchieng Health Centre, Kasy District, Vientiane Province
  - Hinngoon Health Centre, Kasy District, Vientiane Province
  - Kasy District Hospital, Kasy District, Vientiane Province
  - Poonglack Health Centre, Kasy District, Vientiane
  - ThongMeud Health Centre, Kasy District, Vientiane

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for the analysis of the ITCHY trial will be available six months after publication of the primary outcome.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the ITCHY Trial Principle and Associate Investigators must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.

REFERENCES:
- [Derived] Gwee A, Steer A, Phongluxa K, Luangphaxay C, Senggnam K, Philavanh A, Lei A, Martinez A, Huang S, McWhinney B, Ungerer J, Duffull S, Yang W, Zhu X, Coghlan B. Ivermectin therapy for young children with scabies infection: a multicentre phase 2 non-randomized trial. Lancet Reg Health West Pac. 2024 Jul 13;49:101144. doi: 10.1016/j.lanwpc.2024.101144. eCollection 2024 Aug. PMID 39109221